CLINICAL TRIAL: NCT00924872
Title: Power Mobility Training for Persons With Stroke: A Randomized Control Trial
Brief Title: Power Mobility Training for Persons With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Lee Kirby, Attending Staff Physician, Department of Medicine, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDHA-RS-2008-45
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Stroke; Mobility
Keywords: stroke; power wheelchair skills; training; safety
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): receive wheelchair skills training
  Interventions: Other: wheelchair skills training
- control (No Intervention): no formalized wheelchair skills training provided

INTERVENTIONS:
Other: wheelchair skills training — Five 30-minute training sessions, at a target frequency of 3-5 sessions per week, aimed at improving their power wheelchair skills.
  Other Names: WSP
  Arms: intervention

SUMMARY:
To test the hypothesis that persons with stroke can safely and effectively learn to use power mobility devices. The primary objective of this project is to test the hypothesis that, with formal wheelchair skills training, people who have had a stroke and have been prescribed a power wheelchair will have a larger improvement in performance and safety scores on the wheelchair skills test than people who have not received wheelchair skills training.

ELIGIBILITY:
Inclusion Criteria:

* be an inpatient at the Nova Scotia Rehabilitation Centre with a primary diagnosis of stroke within the previous 6 months;
* be competent to provide informed consent;
* have permission of the attending physician to participate;
* require no more than minimal assistance for verbal/non-verbal communication and auditory comprehension as evaluated by a therapist or by chart review of the baseline CIHI evaluation;27
* be able to attend during a 20-minute therapy session as evaluated by the occupational or physical therapist;
* use a manual wheelchair for at least 1 hour per day;
* be able to be safely seated in the power wheelchair that we will be using for the study;
* have no significant visual impairment (such that a subject would be unable to see barriers) as evaluated by his/her therapist based on his/her performance during functional tasks;
* Not currently be using a power wheelchair
* have no physical or mental health condition (as determined by the health-care team) that would make participation dangerous.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Wheelchair skills test - power mobility version | Pre and post intervention, 3 weeks

SECONDARY OUTCOMES:
questionnaire | post intervention (3 weeks), 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lee Kirby, MD, Principal Investigator — Capital Distric Health Authority, Dalhousie University
Locations (1):
- Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- See also: information about wheelchair skills program: training and testing — http://www.wheelchairskillsprogram.ca/